CLINICAL TRIAL: NCT02188355
Title: Prospective, Single Arm, Multi-centre, Observational Registry to Further Validate Safety and Efficacy of the Ultimaster Des System in Unselected Patients Representing Everyday Clinical Practice
Brief Title: Prospective, Single-arm, Multi Centre Observations Ultimaster Des Registry
Acronym: e-Ultimaster
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: T123E2
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease
Keywords: Ultimaster; registry; DES; DAPT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The e-Ultimaster will further validate the safety and efficacy of Ultimaster DES system in unselected patients representing everyday clinical practice. Also the study will assess the impact of non-compliance with dual antiplatelet therapy, one month after stent implementation (frequently observed in every day clinical practice), on stent thrombosis.

DETAILED DESCRIPTION:
All consecutive patients suitable for treatment with DES according to hospital routine practice in centres across the world that agree to participate in the e-ULTIMASTER registry will be treated with Ultimaster DES.

Secondary objectives Evaluation of worldwide utilization of DES, Detection of rare events in representative patient population, identification of predictors of major advers events, assessment of radial access site utilization and its impact on bleeding and vascular complications, assessment of procedural particularities and patients pathology in wide geographic area, assessment of duration and type of DAPT, assesment of the performace of Ultimaster DES is patients lesions subsets, assessment of possible benefits of biodegradable polymer in lager complex patiets/lesions subset and assessment of sirolimus efficacy in different races.

Data will be collected in a e-CRF and online monitoring will be done. Audits will be allowed by sponsor or qualified designees.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* eligible for percutaneous coronary intervention using DES (and RVD matches available Ultimaster DES sizes)
* informed about the nature of the study and agreess to its provisionss and has provided written informed consent as approved by the Institutional Review Board / Ethics committee of the respective clinical site, wherever such requirement exists.

Exclusion Criteria:

* following instruction for use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient 18 years or older eligible for percutaneous coronary intervention using DES
Sampling Method: Probability Sample
Enrollment: 37000 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
TLF | 1 year
  Target Lesion Failure defined as a composite of cardiac death, target vessel related myocardial infarction (MI) and clinically drive target lesion revascularization (TLR) at 1 year.

SECONDARY OUTCOMES:
success endpoints | 3 months and 1 year
  Procedural success and Device success
safety endpoints | 3months and 1 year
  cardiac death / mi (peri and post procedural) stent thrombosis (according to ARC definitions) acute/subacute/late primary/secondary Composite endpoint of cardiac death and post procedural MI Composite endpoint of cardiac death , post procedural MI and stent thrombosis rate during the course of DAPT versus the same events after cessaton of DAPT Major vascular and bleeding complications
efficacy and patient oriented (composite) endpoints | 3months and 1 year
  TLR rate (re-pci/CABG) TLF rate Target Vessel Failure rate (TVF) defined as target vessel revascularization target vessel related q-wave or non q-wave myocardial infarction, or cardiax death that could ot be clearly attributed to a veessl other than the target vessel Patient oriented composite endpoint (POCE) defined as any cause of mortality, mi (q-wave and non qwave) or any TVR

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Borovicanin, MD, Study Director — Terumo Europe
Locations (462):
- Argentina (8):
  - Fundación Favaloro, Buenos Aires
  - Hospital San Juan de Dios, Buenos Aires
  - Hospital Universitario Austral, Buenos Aires
  - Instituto Cardiovascular de Buenos Aires, CABA - Buenos Aires
  - Clinica Centro Médico Privado Junin, Junín
  - Clinica Monte Grande, Monte Grande
  - Instituto Cardiovascular de Rosario, Rosario
  - Sanatorio San Miguel, San Miguel
- Armenia (6):
  - Medical center Gyumri CJSC, Gyumri
  - "QANCOR" cardiovascular MC LLC, Yerevan
  - Astghik Medical Center (Natali Farm), Yerevan
  - QANCOR Cardiovascular MC LLC, Yerevan
  - Republican Medical Center Armenia CJSC, Yerevan
  - Yerevan State medical University Hospital, Yerevan
- Austria (5):
  - Medizinische Universität Graz, Graz
  - AKh Linz, Linz
  - Hanusch Krankenhaus der Wiener Gebietskrankenkasse, Vienna
  - Krankenanstalt Rudolfstiftung der Stadt Wien, Vienna
  - Vienna General Hospital, Vienna
- National Heart Foundation Hospital and Research Institute, Dhākuli, Bangladesh
- Belarus (2):
  - City Clinical Emergency Hospital, Minsk
  - RSPC, Minsk
- Belgium (12):
  - OLVZ Aalst, Onze Lieve Vrouw Ziekenhuis vzw-Campus Aalst, Aalst
  - Olvz Aalst, Aalst
  - Imelda Ziekenhuis - Bonheiden, Bonheiden
  - Imelda Ziekenhuis, Bonheiden
  - Cliniques Saint-Luc, Brussels
  - CHU Charleroi, Charleroi
  - AZ Sint Lucas, Ghent
  - Epicura-Hornu, Hornu
  - Jan Yperman Ziekenhuis, Ieper
  - CHR de la Citadelle, Liège
  - Hôpital Ambroise Paré de Mons, Mons
  - CHU UCL Mont Godinne Namur, Yvoir
- Brazil (11):
  - Hospital Felicio Rocho, Belo Horizonte
  - Unimed Joinville, Joinville
  - Hospital Monte Sinai, Juiz de Fora
  - UNICOR, Linhares
  - Paraná Medical Research Center, Maringá
  - Eurolatino Natal Medical Research, Natal
  - Hospital São Vicente de Paulo, Passo Fundo
  - Hospital Moinhos de Vento, Porto Alegre
  - Hospital e Maternidade Dr. Christóvão da Gama, Santo André
  - Beneficência Portuguesa de São Paulo, São Paulo
  - Hospital Santa Cruz, São Paulo
- Bulgaria (19):
  - "Mhat Puls" Ad, Blagoevgrad
  - City clinic Burgas, Burgas
  - MBAL Haskovo AD, Haskovo
  - Cardiolife-Lovech, Lovech
  - Mbal Montana City Clinic Sveti Georgi, Montana
  - MBAL St. Karidad, Plovdiv
  - MHAT Plovdiv, Plovdiv
  - University Hospital Sveti Georgi, Plovdiv
  - City clinic University Multi-Profile Hospital for Acute Care,Sofia, Sofia
  - MBAZ-II-Sofia, Sofia
  - MHATEM N.I.Pirogov, Sofia
  - National Heart Hospital, Sofia
  - Tokuda Hospital, Sofia
  - UMHAT Alexandrovska, Sofia
  - UMHAT St.Ekaterina, Sofia
  - Trakiya Hospital, Stara Zagora
  - Umbal Stojan Kirkovich, Stara Zagora
  - Specialized Cardiology Hospital for Active Treatment, Varna
  - MBAL Sveta Petka Vidin, Vidin
- Chile (8):
  - Hospital Antofagasta, Antofagasta
  - Hospital Guillermo Grant Benavente, Concepción
  - Hospital Regional Puerto Montt, Port Montt
  - Clinica Bicentenario, Region Metropolitana
  - Clinica Santa Maria, Santiago
  - Hospital San Borja Arriaran, Santiago
  - Hospital San Juan de Dios, Santiago
  - Hospital Van Buren, Valparaíso
- Colombia (5):
  - Clinica Marly, Bogotá
  - Clinica Shaio, Bogotá
  - Fundación Cardiovascular de Colombia, Bucaramanga
  - Instituto del corazón de Bucaramanga, Bucaramanga
  - Centro Cardiovascular de Caldas, Manizales
- Czechia (5):
  - FNKV, Prague, Srobarova
  - Fakultni nemocnice u svate Anny v Brne, Brno
  - Karlovarská Krajská nemocnice, Karlovy Vary
  - Kardiologie na Bulovce, Prague
  - Krajska nemocnice t. Bati, Zlín
- Egypt (15):
  - Police Hospital, Alexandria
  - Al Hayat Hospital, Cairo
  - Al Nakheel Hospital, Cairo
  - Dr Ahmed Abdel Aziz Multicenter, Cairo
  - Dr Hisham Ammar Multicenter, Cairo
  - Dr Hussien Heshmat - As Salam International Hospital, Cairo
  - Dr. Tarek Rashid, Cairo
  - Dr.Hazem Al Guindi, Cairo
  - El Marwa Hospital, Cairo
  - Italian Hospital, Cairo
  - Nile Badrawy Hospital, Cairo
  - Sheraton Hospital for Medical Services, Cairo
  - Wadi El Neel Hospital, Cairo
  - Um El Korra Hospital, El Gharbeya
  - L-Fouad Cardiac Center, Menofia
- Estonia (2):
  - East-Tallinn Central Hospital, Tallinn
  - North Estonia Medical Center, Tallinn
- France (48):
  - CHU Angers, Angers
  - Hopital Européen de Paris La Roseraie, Aubervilliers
  - Clinique Rhône Durance, Avignon
  - GCS Cardiologique de Bayonne, Bayonne
  - Clinique St Augustin Bordeaux-Centre d'exploration-chirurgie, Bordeaux
  - CHU Caen, Caen
  - Hopital Privé Saint Martin, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Pôle Santé République Clermont Ferrand, Clermont-Ferrand
  - Hopital Albert Schweitzer GHCA Colmar, Colmar
  - CH Sud Francilien, Corbeil-Essonnes
  - Clinique de Fontaine, Dijon
  - Groupement mutualiste de Grenoble, Grenoble
  - CH Haguenau, Haguenau
  - CH de Marne la Vallée, Jossigny
  - CHD Vendée La Roche sur Yon, La Roche-sur-Yon
  - Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle
  - CH Louis Pasteur-Le Coudray, Le Coudray
  - Hopital privé La Louviere-Lille, Lille
  - CH St Joseph St Luc Lyon, Lyon
  - Hopital Privé Jacques Cartier Massy, Massy
  - Clinique du Pont de Chaume Montauban, Montauban
  - Clinique du Milénaire, Montpellier
  - CH Montreuil, Montreuil
  - Clinique Diaconat Fonderie Mulhouse, Mulhouse
  - Clinique Louis Pasteur Essey les Nancy, Nancy
  - Le Confluent Nouvelles Cliniques Nantaises, Nantes
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Polyclinique les Fleurs, Ollioules
  - CHR Orléans, Orléans
  - Groupe Hopitalier Paris Saint Joseph, Paris
  - Centre Hospitalier de Pau, Pau
  - Hopital privé St Martin Pessac (DR Levy), Pessac
  - Hôpital Privé St Martin de Pessac, Pessac
  - CHU de Poitiers, Poitiers
  - CH René Dubos Pontoise, Pontoise
  - CHIC Quimper, Quimper
  - Hopiatl Privé Claude Galien Quincy, Quincy-sous-Sénart
  - Clinique Saint-Laurent Rennes, Rennes
  - Clinique ST Hilaire Rouen, Rouen
  - CH Yves le Foll - Saint Brieuc, Saint-Brieuc
  - Institut Arnault Tzanck St Laurent du Var, Saint-Laurent-du-Var
  - CH La Timone Marseille, Saint-Pierre
  - CH Général de Saint Quentin, Saint-Quentin
  - Nouvel Hopital Civil de Strasbourg, Strasbourg
  - Clinique Saint Joseph, Trélazé
  - CH de Valence, Valence
  - CH Bretagne Atlantique, Vannes
- Georgia (3):
  - Diagnostic Services Ltd. Cardio Clinic, Tbilisi
  - Helsicore Clinic, Tbilisi
  - JoAnn Medical Center, Tbilisi
- Hungary (6):
  - Semmelweis University, Budapest
  - Hospital Pándy Kálmán, Gyula
  - Moritz Kaposi General Hospital, Kaposvár
  - Szatmar-Szabolcs-Bereg county hospital and university teaching hospital, Nyíregyháza
  - Pecs University, Pécs
  - Markusovszky University Teaching Hospital, Szombathely
- Landspitali National University hospital, Reykjavik, Iceland
- India (15):
  - Kamalnayan Bajaj Hospital, Aurangabad
  - MMM, Chennai, Chennai
  - G. Kuppuswamy Naidu Memorial Hospital (GKNM), Coimbatore, Coimbatore
  - Medanta Hospital, Delhi, Delhi
  - Care Hospital, Hyderabad, Hyderabad
  - SMS Hospital, Jaipur, Jaipur
  - BM Birla, Kolkata, Kolkata
  - KMC, Mangalore, Mangalore
  - Fortis Hospital, Mohali, Mohali
  - H.J. Doshi Ghatkopar Hindusabha Hospital, Mumbai
  - Hiranandani Hospital, Mumbai, Mumbai
  - Wockhardt Hospital, Nagpur, Nagpur
  - Maharaja Agrasen Hospital, New Delhi, New Delhi
  - Max Super Speciality Hospital, Saket, Delhi, New Delhi
  - SCTIT, Trivanderum, Trivanderum
- Indonesia (9):
  - Medistra Hospital, Jakarta
  - National Cardiovascular Center Harapan Kita, Jakarta Barat
  - RSUPN Cipto Mangunkusumo, Jakarta Pusat
  - RSUP Fatmawati General Hospital, Jakarta Selatan
  - Binawaluya Cardiac Center, Jakarta Timur
  - Awal Bros Hospital, Makassar
  - Dr. Wahidin Sudirohusodo General Hospital, Makassar
  - Saiful Anwar Hospital, Malang
  - Dr. Soetomo General Hospital, Surabaya
- Ireland (3):
  - Cork University Hospital, Cork
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
- Israel (4):
  - Rambam Medical Center, Haifa
  - Galilee Medical Center, Nahariya
  - Ziv M.C, Safed
  - Assaf Harofeh Medical Center, Tzrifin
- Japan (26):
  - Kansai Rosai Hospital, Amagasaki Hyougo
  - Kokura Memorial Hospital, Fukuoka
  - Iwaki Kyoritsu General Hospital, Fukushima
  - Tokai University Hachiouji Hospital, Hachiōji
  - Hakodate Municipal Hospital, Hakodate Hokkaido
  - Seirei Hamamatsu General Hospital, Hamamatsu
  - Kakogawa East City Hospital, Kakogawa
  - Shonan Kamakura General Hospital, Kanagawa
  - Komaki City Hospital, Komaki Aichi
  - Kyoto Katsura Hospital, Kyoto
  - Gunma Prefectural Cardiovascular Center, Maebashi
  - Mie Heart Center, Mie
  - Osaka General Medical Center, Osaka
  - Sakurabashi Watanabe Hospital, Osaka
  - Saitama Cardiovascular and Respiratory Center, Saitama
  - Mimihara General Hospital, Sakai
  - Osaka Rosai Hospital, Sakai Osaka
  - Sapporo Higashi Tokushukai Hospital, Sapporo Hokkaido
  - Saiseikai Senri Hospital, Suita
  - Okamura Memorial Hospital, Suntougun Shizuoka
  - Higashi Takarazuka Satoh Hospital, Takarazuka Hyougo
  - Kouseikai Takai Hospital, Tennri Nara
  - Saiseikai Yamaguchi General Hospital, Yamaguchi
  - Saiseikai Yokohama City Eastern Hospital, Yokohama
  - Seirei Yokohama Hospital, Yokohama
  - Showa University Fujigaoka Hospital, Yokohama Kanagawa
- Jordan Hospital, Amman, Jordan
- Kazakhstan (16):
  - Aktobe Regional Hospital, Aktobe
  - Medical University Clinic West Kazakhstan, Aktobe
  - Almaty city cardio center, Almaty
  - National Surgery Center Almat, Almaty
  - City Hospital #2, Astana
  - JSC Nat. Scient. Cardiosurgery Ctr., Astana
  - National Scientific Medical Research Center JSC, Astana
  - Karagandy Regional Cardiac Center, Karaganda
  - Regional Cardiosurgery Center, Karaganda
  - Akmola Regional Hospital, Kokshetau
  - Pavlodar Regional Cardiologic center, Pavlodar
  - Cardiology Center Petropavl, Petropavl
  - Rudnyi City Hospital, Rudnyi
  - University Hospital of Semey, Semey
  - Shymkent Regional Cardiology Center, Shymkent
  - Clinical Center of Cardiac Surgery and Transplantation, Taraz
- Sabah Al Ahmad Cardiac Center, Kuwait City, Kuwait
- Lebanon (2):
  - Hopital Abou Jaoudé, Beirut
  - Labib Medical Center, Sidon
- Lithuania (2):
  - LSMU Kauno Klinikos, Kaunas
  - Klaipeda Seamen's Hospital, Klaipėda
- Malaysia (6):
  - Hospital Sultanah Bahiyah, Alor Setar, Kedah
  - Hospital Serdang, Kajang
  - Desa Park City, Kuala Lumpur
  - HSC Medical Center, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - UiTM Sg. Buloh Campus, Sungai Buloh
- Mexico (3):
  - Fray Juan de San Miguel, Michoacán
  - Clinica Hospital San Jose de Navojoa SA de CV, Sonora
  - Hospital Star Médica Merida, Yucatán
- Morocco (4):
  - Clinique Achifaa de Casablanca, Casablanca
  - Clinique Grant Atlas, Marrakesh
  - CLINIQUE INTERNATIONALE de Marrakech, Marrakesh
  - Cherradi_Clinique Agdal, Rabat
- Netherlands (14):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Meander Amersfoort, Amersfoort
  - Rijnstate, Arnhem
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina Hospital, Eindhoven
  - Catharina Ziekenhuis, Eindhoven
  - Scheper Ziekenhuis, Emmen
  - Medisch Spectrum Twente, Enschede
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Maasstad Ziekenhuis, Rotterdam
  - Zorgzaam Ziekenhuis Zeeuws-Vlaanderen, Terneuzen
  - Medisch Centrum Haaglanden, The Hague
  - VieCuri Medical Centre, Venlo
- North Macedonia (2):
  - City General Hospital 8th September Skopje, Skopje
  - University Clinic of Cardiology, Skopje
- Muscat Private Hospital, Muscat, Oman
- Poland (4):
  - Miedziowe Centrum Zdrowia, Lubin
  - Szpital Kliniczny Przemienienia Panskiego UM im. K. Marcinkowskiego w Poznaniu, Poznan
  - Infant Jesus Teaching Hospital, Warsaw
  - Instytut Kardiologii im. Prymasa Tysiąclecia Stefana Kardynała Wyszyńskiego, Warsaw
- Hospital Santa María, Lisbon, Portugal
- Romania (4):
  - Clinicile ICCO, Brasov
  - Centrele de Exelenta ARES, Constanța
  - Spitalul Judetean de Urgenta Sibiu, Sibiu
  - Cordismed SRL, Timișoara
- Saudi Arabia (2):
  - Prince Abdullah Bin Abdulaziz Cardiac Center, North Region Arar KSA
  - Dallah Hospital, Riyadh
- Serbia (6):
  - Cardiology Clinic, Clinical Centre of Serbia, Belgrade
  - Cardiovascular Institute Dedinje, Belgrade
  - CHC Bezanijska kosa, Belgrade
  - KBC Zvezdara, Belgrade
  - Institute of cardiovascular diseases Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
- Stredodlovensky Ustav Srdcovych A Cievnych Chorob, Banská Bystrica, Slovakia
- South Africa (8):
  - Dr JCW Badenhorst - Netcare Unitas Hospital, Centurion
  - Unitas Hospital - Dr. Ebrahim, Centurion
  - Unitas Hospital, Centurion
  - Milpark Hospital, Johannesburg
  - Netcare Union Hospital, Johannesburg
  - Ethekwini Hospital & Heart centre, Newlands
  - Netcare Greenacres Hospital, Port Elizabeth
  - Netcare Unitas Hospital, Pretoria
- Spain (60):
  - Complexo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital San Rafael (La Coruña), A Coruña
  - Hospital general de Albacete, Albacete
  - Hospital General de Alicante, Alicante
  - Hospital Infanta Cristina - Badajoz, Badajoz
  - Hospital G. Trias i Pujol (Badalona), Badalona
  - Hospital de Cruces-Barakaldo, Barakaldo
  - Bellvitge University Hospital, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Sant Pau (Barcelona), Barcelona
  - Hospital V. Hebrón, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Galdakano, Bizkaia
  - Hospital General Universitario de Burgos, Burgos
  - Hospital Santa Lucia de Cartagena, Cartagena
  - Universitario Santa Lucia (Hospital Nostra Señora Rossell) (Cartagena), Cartagena
  - Hospital Santa Lucia de Cartagena, Cartagena (Murcia)
  - Hospital General Castellón, Castellon
  - Hospital San Pedro de Alcantara-Caceres, Cáceres
  - Hospital General Ciudad Real, Ciudad Real
  - Hospital de la Cruz Roja de Córdoba, Córdoba
  - Hospital Reina Sofia de Córdoba, Córdoba
  - Hospital de Galdakao, Galdakao
  - Hospital Cabueñes (Gijón), Gijón
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Juan Ramón Jiménez, Huelva
  - Hosp Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital de León, León
  - Hospital San Pedro (Logroño - La Rioja), Logroño
  - Hospital San Pedro, Logroño
  - Hospital Universitario Lucus Augusti (HULA), Lugo
  - Clinica La Luz, Madrid
  - Clínica San Fransisco de Asis (Madrid), Madrid
  - Hospital 12 Octubre, Madrid
  - Hospital Fundacion Alcorcon, Madrid
  - Hospital La Luz, Madrid
  - Hospital Moncloa (Madrid), Madrid
  - Hospital Moncloa, Madrid
  - Hospital Puerta de Hierro (Madrid), Majadahonda
  - Hospital Manises (Valencia), Manises
  - Hospital de Mérida, Mérida
  - Hospital Virgen Arrixaca (Murcia), Murcia
  - Universitario central de Asturias (Oviedo), Oviedo
  - Universitario central de Asturias, Oviedo
  - Hospital de Navarra, Pamplona
  - San Juan de Alicante, San Juan
  - Hospital de Donostia, San Sebastián
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Marqués de Valdecilla, Santander, Santander
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Virgen De La Salud (Toledo), Toledo
  - Hospital Virgen De La Salud, Toledo
  - Clínico Universitario Valencia, Valencia
  - Instituto Cardiologico Hospital Campo Grande (Valladolid), Valladolid
  - Instituto Cardiologico Hospital Campo Grande, Valladolid
  - Hospital Meixoeiro-MEDTEC (Vigo), Vigo
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital Clínico Lozano Blesa de Zaragoza, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (9):
  - Gavle Sjukhus, Gävle
  - Malarsjukshuet, Malarsjukhuset
  - sjukhuset Orebro, Örebro
  - Universitets Sjukhuset I Örebro, Örebro
  - Skaraborgs sjukhus v Skövde, Skövde
  - Skaraborgs Sjukhus, Skövde
  - Sundvalls Sjukhus, Sundvalls
  - Vastmanlads Sjukhus, Västerås
  - Västmanlads sjukhus Västerås, Västerås
- Switzerland (9):
  - Spital Thurgau AG, Frauenfeld
  - Hopitaux Universitaires de Genève, Geneva
  - Kantonsspital Baselland, Liestal
  - Kantonsspital Luzern, Lucerne
  - Cardiocenter Lugano, Ticino (TI), Lugano
  - Cardiocentro Ticino, Lugano
  - La Tour Hospital, Meyrin Geneva
  - HerzGefässZentrum Zürich, Zurich
  - HerzGefässZentrum, Zurich
- Thailand (9):
  - Paolo Memorial Hospital Phaholyothin, Bangkok
  - Police General Hospital, Bangkok
  - Ramkhamhaeng Hospital, Bangkok
  - HRH Princess Maha Chakri Siridhorn Medical Center, Nakhon Navok
  - HRH Princess Maha Chakri Sirindhorn Medical Center (Nakornayok), Nakhon Navok
  - Central Chest Institute of Thailand, Nonthaburi
  - Phatara Thonburi Hospital, Pathum Thani
  - Udonthani Hospital, Udon Thani
  - Udonthani HP., Udon Thani
- Tunisia (16):
  - Clinique Hannibal Lac 2_Dr. Mohamed Drissa, El Mourouj
  - Clinique Générale et Cardiovasculaire de Tunis_Dr. Sami Bouziri, La Marsa
  - Bassatine Clinic_Dr. Elyes Kharrat, Sfax
  - Polyclinique Bassatine Cite gardin Sfax_Dr. Zeineb Grati Guermazi, Sfax
  - Polyclinique El Bassatine SFAX_Dr. Sami Fourati, Sfax
  - Polyclinique El bassatine_Dr. Mohamed Najeh Abid, Sfax
  - Polyclinique El Bassatine_Dr. Ridha Ennouri, Sfax
  - Centre Urbain Nord_Dr. Salem Abdessalem, Tunis
  - Clinique Cartagène_Dr. Dhaker Lahidheb, Tunis
  - Clinique Général et Cardiovasculaire de Tunis_Dr. Saloua Trabelsi, Tunis
  - Clinique Générale et Cardiovasculaire de Tunis_Dr. Saloua TRABELSI, Tunis
  - Clinique Hannibal Lac 2_Gharbi Mostari, Tunis
  - Clinique Montplaisir_Dr. Badi Darghouth, Tunis
  - HU Mohamed Taher El Maâmouri, Tunis
  - Policlinique Taoufik_Jamel Langar, Tunis
  - Soukra Medical_Dr. Ben Chedli Tarek, Tunis
- Ukraine (9):
  - Heart Institute, Kiev
  - Institute of Heart (Ministry of Health), Kiev
  - NAMS Amosov | Emergency Endovascular Surgery department, Kiev
  - NAMS Amosov | X-Ray diagnostics and invasive cardiology department, Kiev
  - National Institute of Cardiovascular Surgery NAMS, Kiev
  - National Institute of Surgery and Transplantology NAMS, Kiev
  - S.P.M.C. of Pediatric Cardiology and Cardiac Surgery, Kiev
  - Strazhesko Institute of Cardiology (National Scientific Centre), Kiev
  - Government institution Regional centre of cardiac and vessel disease, Zaporizhzhya
- United Arab Emirates (10):
  - Al Noor Hospital-Airport Rd., Abu Dhabi
  - LifeCare Hospital, Abu Dhabi
  - Al Zahra Private hospital, Dubai, Dubai
  - Belhoul Speciality Hospital, Dubai
  - Dr. Sulaiman Al Habib Hospital, Dubai
  - Dubai Hospital, Dubai
  - Iranian hospital, Dubai
  - Prime Hospital, Dubai
  - Rashid Hospital, Dubai
  - Al Qassimi Hopsital, Sharjah city
- United Kingdom (46):
  - Royal Brompton and Harefield, Chelsea, London
  - Essex Cardiothoracic centre, Basildon
  - Royal United Hospital, Bath, Bath
  - Bedford Hospital, Bedford
  - Queen Elizabeth Hospital, Birmingham
  - Sandwell and West Birmingham Hospitals, Birmingham
  - Royal Blackburn Hospital, Blackburn
  - Blackpool Victoria Hospital, Blackpool
  - Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth
  - Bradford teaching hospitals, Bradford
  - Royal Sussex Hospital, Brighton, Brighton
  - University Hospital Wales, Cardiff
  - Croydon University Hospital, Croydon
  - Royal Derby Hospital, Derby
  - Dorset County Hospital, Dorchester
  - Eastbourne and Conquest Hospitals, Eastbourne
  - Freeman Hospital, Freeman
  - Buckinghamshire, Wycombe, High Wycombe
  - West Middlesex Hospital, Isleworth
  - Kettering General Hospital, Kettering
  - University Hospitals of Leicester, Leicester
  - Lincoln County Hospital, Lincoln
  - Royal Free Hospital, London
  - The Royal Free Hospital, London
  - University Hospital of South Manchester, Manchester
  - James Cook University Hospital, Middlesbrough
  - Wolverhampton, New Cross
  - Royal Gwent Hospital, Newport, Newport
  - Northwick Park Hospital, Northwick Park
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham University Hospitals - Queen's Medical Centre, Nottingham
  - Queens medical center Nottingham, Nottingham
  - Bircham Park Offices Plymouth, Plymouth
  - Plymouth Hospital, Plymouth
  - Royal Berkshire, Reading
  - Tunbridge Wells Hospital, Royal Tunbridge Wells
  - Salisbury District Hospital, Salisbury
  - Sheffield teaching hospital, Sheffield
  - Lister Hospital, Stevenage, Stevenage
  - Royal Stoke University Hospital, Stoke-on-Trent
  - King's Mill Hospital, Sutton in Ashfield
  - Royal Cornwall Hospitals, Truro
  - Coventry and Warwickshire, Walsgrave on Sowe
  - Wrightington Hospital, Wigan
  - Worcestershire Acute Hospitals, Worcestershire
  - Worthing Hospital, West Sussex, Worthing
- Republic Specialized Center of Surgery, Tashkent, Uzbekistan
- Thong Nhat Hospital, Hò Chi Minh City, Vietnam

REFERENCES:
- [Derived] Mamas MA, Roffi M, Frobert O, Chieffo A, Beneduce A, Matetic A, Tonino PAL, Paunovic D, Jacobs L, Debrus R, El Aissaoui J, van Leeuwen F, Kontopantelis E. Predicting target lesion failure following percutaneous coronary intervention through machine learning risk assessment models. Eur Heart J Digit Health. 2023 Aug 31;4(6):433-443. doi: 10.1093/ehjdh/ztad051. eCollection 2023 Dec. PMID 38045434
- [Derived] Kobo O, Saada M, von Birgelen C, Tonino PAL, Iniguez-Romo A, Frobert O, Halabi M, Oemrawsingh RM, Polad J, IJsselmuiden AJJ, Roffi M, Aminian A, Mamas MA, Roguin A. Impact of multisite artery disease on clinical outcomes after percutaneous coronary intervention: an analysis from the e-Ultimaster registry. Eur Heart J Qual Care Clin Outcomes. 2023 Jun 21;9(4):417-426. doi: 10.1093/ehjqcco/qcac043. PMID 35876646